CLINICAL TRIAL: NCT02888470
Title: Administration of Amino-glycoside in ICU Patients : Clinical Practices in 2013
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 13 10 02
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of the study is to estimate the proportion of intensive care unit patients receiving current aminoglycosides dosing regimens as part of their antibiotic therapy and achieving the recommended maximal plasma concentration (Cmax) after the first and subsequent aminoglycoside doses.

DETAILED DESCRIPTION:
Aminoglycosides are often prescribed as part of empirical therapy for severe sepsis and septic shock, especially when Gram-negative bacteria are suspected. From a pharmacodynamic perspective, the ratio between the maximal plasma concentration (Cmax) and the minimum inhibitory concentration (MIC) of the infecting pathogen (Cmax/MIC) is considered as the best index of bacterial killing for aminoglycosides. In 2011, French guidelines on aminoglycoside use recommend a targeted Cmax of 30-40 mg/L for gentamicin and 60-80 mg/L for amikacin. However, these recommended plasma levels may not be achieved in high risk patients such as ICU patients. Many factors can influence the pharmacokinetics of antimicrobial drugs in critically ill patients. Indeed, alterations in the volume of distribution, plasma albumin concentration, increased cardiac output, increased blood volume, and paradoxical renal and hepatic clearance increase can be observed in the early stage of severe sepsis and are frequently observed in ICU patients. Previous studies have reported low aminoglycoside plasma concentrations in the early phase of therapy in ICU patients. However, data for the subsequent doses of aminoglycosides were not available. Therefore, to address this lack of data, an observational study is performed to describe the proportion of ICU patients achieving targeted aminoglycoside Cmax after the first and subsequent aminoglycoside doses using conventional dosing regimens.

Aminoglycoside agents are given in combination with broad-spectrum antibiotics according to the suspected pathogens and to local clinical practice. A once-daily dosing regimen based on the French guidelines is used: ≥15 mg/kg for amikacin and ≥3 mg/kg for gentamicin based on actual weight at admission. For obese patients,the weight used for dosing is left to the physician's discretion.All aminoglycosides are given as a 30-min i.v. infusion in glucose 5% solution. The timing of Cmax sampling is 30 min after the end of initial infusion. When subsequent doses of aminoglycoside were recommended as part of the patient's treatment plan, trough plasma concentrations (taken at 16-24 h post-infusion) (Cmin) and Cmax were collected as part of routine practice.The targeted concentrations for amikacin and gentamicin are as follows: amikacin, Cmax ≥60 mg/L and Cmin <2.5 mg/L; and gentamicin, Cmax ≥30 mg/L and Cmin <0.5 mg/L.The following data are collected:•demographic characteristics: age, sex, and height , weight and body mass index (BMI);•medical history, initial reason for ICU admission and Simplified Acute Physiology Score II (SAPS II) at ICU admission;•clinical parameters: urine output; the Sequential Organ Failure Assessment (SOFA) score and the Acute Kidney Injury Network (AKIN) score are calculated daily from the initiation of aminoglycoside therapy;•presence of renal replacement therapy (RRT);•co-prescription of nephrotoxic agents (e.g. glycopeptides, diuretics);•biological parameters: serum creatinine concentration, hepaticf unction (serum total bilirubin and transaminase) and platelets that are daily measured in routine practice;•type of infection and anti-infective therapy and microbiological cultures collected. Amikacin and gentamicin concentrations are measured using automated immunoassays(Roche Diagnostics GmbH, Mannheim, Germany) on a COBAS®C System.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* indication of aminogycoside therapy for a current infectious episode

Exclusion Criteria:

* <18years
* allergy to aminoglycosides
* patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ICU patients with indication of aminoglycosides (gentamicin, tobramycin or amikacin) for a current infectious episode
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Achievement of the recommended Cmax after the first and subsequent aminoglycoside doses. | 7 days